CLINICAL TRIAL: NCT06290492
Title: Clinical Efficacy and Mechanism of High Definition tDCS Based on dmPFC in the Intervention of Chronic Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WANG KAI (Other)
Responsible Party: Sponsor-Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tDCS-insomnia
Record Dates: First submitted 2023-12-28; First posted 2024-03-04 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Chronic Insomnia; Transcranial Direct Current Stimulation
Keywords: Chronic Insomnia; HD-tDCS
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- real stimulation (Active Comparator): Participants will receive active HD-tDCS daily for 10 consecutive days. The anode electrode was placed on the DMPFC (Fz) surrounded by four cathodes with a 1cm diameter (FPz, F3, Cz, and F4). The stimulation direct current magnitude was set at 2 mA with a 30-s immediate decline at the beginning and end of each phase.
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Sham Comparator): In the sham intervention phase, the sensation was simulated by applying a 30-s rising current until 2 mA was reached, with a 30-s immediate decline at the beginning and end of each phase.
  Interventions: Device: sham transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, direct current applied directly to the head through scalp electrodes
  Arms: real stimulation
Device: sham transcranial direct current stimulation — Sham tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of transcranial direct current stimulation (tDCS) on subjective and objective insomnia symptoms and daytime function of chronic insomnia patients.

DETAILED DESCRIPTION:
Fifty patients with chronic insomnia disorder diagnosed by the Diagnostic Criteria and Treatment Guidelines for Adult Insomnia (2017) were recruited from the first affiliated Hospital of Anhui Medical University. After meeting the inclusion criteria and obtaining informed consent, each participant will complete the subjective measures consisting of sleep questionnaires, polysomnography (PSG) and tDCS treatment conducted by trained researchers at the Neurology Department of Anhui Medical University. All the participants were randomized (1:1) to receive "active" or "sham" treatment protocol. The anode electrode was placed on the DMPFC (Fz) surrounded by four cathodes with a 1cm diameter (FPz, F3, Cz, and F4). Each participant received 30 min of tDCS stimulation once daily for 10 consecutive days. The stimulation direct current magnitude was set at 2 mA in the active group. In the sham intervention phase, the sensation was simulated by applying a 30s rising current until 2 mA was reached, with a 30s immediate decline at the beginning and end of each phase.

At the beginning and after a 10-day intervention, subjective measures consisting of sleep questionnaires, including the Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI), were assessed. The Flinders Fatigue Scale (FFS) and the Epworth Sleepiness Scale (ESS) were used to assess daytime sleepiness. Additionally, the HAMA and HAMD were used synchronously for emotional assessment. Afterwards, they were unblinded by the study coordinator.

ELIGIBILITY:
Inclusion Criteria:

1. age between 15 and 65 years,
2. diagnosed with chronic insomnia based on the Diagnostic Criteria and Treatment Guidelines for Adult Insomnia (2017),
3. no previous application of any insomnia pharmacological therapy for at least one week before baseline visit.

Exclusion Criteria:

1. diagnosis of other sleep disorders, such as sleep apnoea-hypopnoea syndrome, REM behaviour disorder, and restless legs syndrome,
2. history of head trauma or presence of serious organic diseases,
3. presence of comorbid anxiety or depression, as assessed by a Hamilton Anxiety Scale [HAMA] score of 17 or Hamilton Depression Scale [HAMD] score of 14.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
subjective sleep quality assessed by the PSQI | before and after 10-day intervention
  The Pittsburgh Sleep Quality Index (PSQI) consist of 18 items divided into 7 dimensions, such as sleep duration, sleep efficiency, sleep disorders and daytime dysfunction. The PSQI total score ranges from 0 to 21, the higher the score indicates the more worse sleep quality.
subjective sleep quality assessed by the ISI | before and after 10-day intervention
  The Insomnia Severity Index (ISI) is a 7-item scale to measure insomnia symptoms, where each item is rated on a scale from 0 to 4. The ISI total score ranges from 0 to 28, The higher the score indicates the more worse sleep quality.
daytime sleepiness assessed by the FFS | before and after 10-day intervention
  the Fatigue Severity Scale (FFS) is a 7-item scale to measure daytime sleepiness, where each item is rated on a scale from 0 to 3. The FFS total score ranges from 0 to 31, the higher the score indicates the more serious daytime sleepiness.
daytime sleepiness assessed by the ESS | before and after 10-day intervention
  The Epworth Sleepiness Scale (ESS) is a 8-item scale to measure daytime sleepiness, where each item is rated on a scale from 0 to 3. The ESS total score ranges from 0 to 23, the higher the score indicates the more serious daytime sleepiness.
objective sleep quality assessed by the PSG | before and after 10-day intervention
  the change of objective sleep quality assessed by polysomnography(PSG) will constitute the major research outcome measure, to assess response to tDCS. Recorded details included data on SOL(sleep onset latency), TST(total sleep time), WASO(wake after sleep onset), EF(sleep Efficiency), and percentages of slow-wave sleep, stage 2 sleep, stage 1 sleep, and REM sleep.

SECONDARY OUTCOMES:
emotional symptoms assessed by the HAMA | before and after 10-day intervention
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
emotional symptoms assessed by the HAMD | before and after 10-day intervention
  The HAMD is a clinic ian-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China